CLINICAL TRIAL: NCT02822196
Title: Effectiveness of Serratus Anterior Muscle Plane Block With Thoracic Paravertebral Block For Unilateral Mastectomies
Brief Title: Serratus Anterior Muscle Plane Block vsThoracic Paravertebral Block For Unilateral Mastectomies
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Critical study personnel left the institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Sara R Guzman-Reyes, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-16-0467
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Mastectomy; Regional Anesthesia; Post Operative Pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative | interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus Anterior Muscle Plane Block (Experimental): The US probe will be placed in the mid-axillary line at the level of the 5th intercostal space. The latissimus dorsi, teres major and serratus muscles will be identified. Using in-plane approach, the block needle (22 G, 50 mm) will be inserted until the tip is visualized between the serratus anterior muscle and the intercostal muscles. As an extra reference point thoracodorsal artery will be used which aids in the identification of the plane superficial to the serratus muscle. After negative aspiration of blood, local anesthetic (20 ml of 0.25 % bupivacaine) will be injected and visualized in real-time.
  Interventions: Drug: Bupivacaine
- Thoracic Paravertebral Block (Active Comparator): The spinous processes of T1- T5 will be identified and at parasagittal plan at 2.5 cm, skin wheel will be raised using 1% lidocaine. A 20-gauge, bevel needle will be advanced until the transverse process is located. The depth from skin to transverse process will be marked/identified by needle marking. The needle will be withdrawn 1-2 cm and angled down.The needle will be re-advanced 1cm past the initial marking. After negative aspiration, 4-5 ml of 0.25% bupivacaine will be slowly injected. The same procedure will be repeated at each level from T2 to T6 ensuring total dose of bupivacaine does not exceed the maximum dose recommended.
  Interventions: Drug: Lidocaine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Lidocaine — Local Anesthesia using 1% Lidocaine
  Other Names: 1% Lidocaine
  Arms: Thoracic Paravertebral Block
Drug: Bupivacaine — Local Anesthesia using 0.25% Bupivacaine
  Other Names: 0.25% Bupivacaine

SUMMARY:
HYPOTHESIS

Serratus Anterior Muscle Plane Block (SPB) is as effective as thoracic paravertebral block (PVB) for acute pain control after unilateral mastectomies.

SPECIFIC AIMS

Primary aim: To evaluate the efficacy of SPB block vs thoracic PVB for acute pain control in patients undergoing unilateral mastectomy

Secondary aim To compare the onset and duration of block and dermatomes blocked in both groups To compare the need of post-operative rescue analgesia in both groups. To compare the development of chronic incisional pain in both groups Functional outcome with respect to daily activities.

DETAILED DESCRIPTION:
RESEARCH STRATEGY

1. Background

   Breast cancer is a potentially deadly disease affecting one in eight women. [1] Majority of them undergo mastectomies along with different modalities of treatment like chemotherapy, radiotherapy and hormonal treatments.

   Since mastectomy is the main and most commonly preferred treatment for breast cancer surgery, it raises the focus on the most frequently studied complication that is persistent pain following surgery [8, 9] The incidence of pain syndrome six months post-breast cancer surgical treatment was 52.9%.[7] A multivariate analysis of the presence of chronic pain in breast cancer survivors revealed risk factors including more invasive surgery, radiation therapy after surgery, and clinically meaningful acute postoperative pain. Each risk factor independently predicted more intense chronic pain at three months after surgery. [8] A 20% prevalence rate of the Post Mastectomy Pain syndrome was found. Women experiencing the syndrome reported chronic, stable pain of long duration that began shortly after surgery. [10] The syndrome is important to recognize because of how debilitating the pain can be. Studies have indicated that post mastectomy pain interferes with activities of daily living like driving, taking care of the children, leisure time, and sex, all of which result in poor quality of life. It was also noted that in women who survived treatment of breast cancer, chronic pain often caused mood changes, difficulty at work, and reduction of physical activities. This was especially noted in those women whose pain spreads to other areas of the body. [14]

   There are various anesthetic techniques available for management of mastectomies. The effectiveness of each technique is widely studied regarding pain control, requirement of rescue analgesia, side effects, post-operative hospital stay and development of persistent pain following breast cancer surgical treatment. Belzarena SD et al compared the effectiveness of thoracic epidural block and general anesthesia for oncologic mastectomy. Patients were divided in two groups in which they either received GA or thoracic epidural anesthesia as primary anesthetic. [10] The results showed that the quality of postoperative analgesia was better in the epidural group, which also presented with lower consumption of analgesics. The length hospitalization in this group was also lower. They concluded that an epidural block had some advantages when compared with general anesthesia and can be considered an anesthesia option in oncologic mastectomies with axillary lymph node dissection.

   Newer regional anesthesia techniques have been developed to improve pain control and patient satisfaction. These includes epidural blocks (thoracic and cervical), single injection thoracic PVB and intercostal nerve blocks. PVB during breast cancer surgery have been reported to decrease acute pain and opioid consumption immediately following surgery in multiple randomized clinical trials [4, 5, 6] and were superior over epidural blocks due to lower complication rate. A thoracic PVB is a well-established anesthetic technique and has been proven to be safe for mastectomies.

   The most recent advancement in anesthetic techniques for mastectomies is the SPB. The SPB is a novel technique first described by Fajardo et al in 2012 [2]. A single injection blocks many dermatomes at once. This technique could be an effective alternative to PVB or thoracic epidurals, because it is considered more feasible, safe than thoracic epidurals and results in a lower complication rate. But there are very few long term randomized studies to prove the efficacy of SPB.

   R. Blanco et al studied this novel ultrasound-guided regional anesthetic technique to provide analgesia following surgery on the thoracic wall in four volunteers. All volunteers reported an effective block that provided long-lasting paresthesia (750-840 min). There were no side-effects noted in this initial descriptive study. They have suggested to confirm these preliminary results in a large clinical trial.[12] Currently only a single major clinical trial comparing the effectiveness of SPB and PVB for Breast Cancer Resections is being conducted by Ghada M N Bashandy, National Cancer Institute, Egypt. [13]
2. Protocol/Experimental Design/Flowchart/Primary and Secondary End Points

   Criteria

   Ages Eligible for Study: 18 Years to 80 Years Genders Eligible for Study: Female No. of subjects in each group: 50. (Total = 100)

   Informed consent for the procedure will be taken. Patients will be educated on the use of the visual analogue scale (VAS) to evaluate their pain level and a printed copy of the VAS scoring will be provided to take home. After the completion of preoperative assessment by the OR nurse, the patients will be randomized to either SPB group or PVB group. The block will be performed pre operatively. To reduce patient anxiety and improve comfort, midazolam 0.02mg/kg IV will be given except in patients > 70 years of age. Standard ASA monitors were applied including pulse oximetry, noninvasive blood pressure, and electrocardiogram.

   Procedure: Serratus Anterior Muscle Plane block (SPB)

   The US probe will be placed in the mid-axillary line at the level of the 5th intercostal space. The latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscles (deep and inferior) will be identified. Using in-plane approach, the block needle (22 G, 50 mm) will be inserted until the tip is visualized between the serratus anterior muscle and the intercostal muscles. As an extra reference point thoracodorsal artery will be used which aids in the identification of the plane superficial to the serratus muscle. After negative aspiration of blood, local anesthetic (20 ml of 0.25 % bupivacaine) will be injected and visualized in real-time. [11]

   Procedure: Paravertebral Block (PVB)

   Patients will be placed in the sitting position, leaning forward. After skin disinfection using chlorhexidine solution, target spinous processes of T1- T5 will be identified and at parasagittal plan at 2.5 cm, skin wheel will be raised using 1% lidocaine. A 20-gauge, bevel needle will be advanced until the transverse process is located. The depth from skin to transverse process will be marked/identified by needle marking. The needle will be withdrawn 1-2 cm and angled down (walked off the transverse process). The needle will be re-advanced 1cm past the initial marking. After negative aspiration, 4-5 ml of 0.25% bupivacaine will be slowly injected. The same procedure will be repeated at each level from T2 to T6 ensuring total dose of bupivacaine does not exceed the maximum dose recommended. [13]

   After the block is performed, all subjects will receive induction of general anesthesia with fentanyl 1-2 mcg/kg, propofol 1-2 mg/kg and suxamethonium 1 mg/kg. After induction the trachea will be intubated with 7.0 mm ID endotracheal tube. For analgesia all patients will receive 1 gm of intravenous acetaminophen. Anesthesia will be maintained with sevoflurane with oxygen and air. To minimize PONV, every patient will receive ondansetron 4mg at the end of the surgery. Fentanyl 25 mcg boluses will be used as rescue analgesia intra operatively. When extubation criteria have been met the trachea will be extubated and the patient will be taken to PACU.

   PACU phase I For VAS >6, 0.5 mg intravenous hydromorphone every 10 min up to 2 mg as a rescue analgesia For VAS </=6, patient will be given tramadol 100 mg.

   PACU phase II Prior to discharge all patients will receive tramadol 50mg if they have not required pain medication in phase I.

   At discharge, all patients will be prescribed Norco (7.5/325) every 4 hours prn for VAS>4.

   Reinforcement of previous education on VAS scoring will be done as part of discharge instructions by the discharge nurse.

   The following parameters will be recorded in each group.
   * Duration of block analgesia - time to peak of pain/return of sensation after surgery will be recorded
   * Dermatomal distribution of sensory loss obtained after block tested with ice.
   * Assessment of static and dynamic VAS scores at 0 (on arrival to PACU), 6, 12, 24 and 48 hours, 3 months and 6 months after surgery and additional set of questions to assess neuropathic pain. ( painDETECT)
   * Time for 1st rescue analgesia
   * Total dose of rescue analgesia received during the first 24 and 48 hrs
3. Sample size and statistical analysis

Statistical analysis plan StatistiCall will create the randomization list by using the software ClinStat (from St. George's Hospital Medical School, Version dated 08.05.96). The treatment will be named 1 for SPB Block, 2 for PVB block for both parts of the study in the list. Block randomization in X blocks of X patients will be used.

Since there is no valid data comparing the 2 blocks, we are unable to construct a realistic power analysis as the hypothesis of difference between the 2 procedures are potentially minimal and not yet statistically proven. Therefore, this initial investigation in 100 subjects is clinically and logistically feasible and analysis will provide statistical guidance to any necessary additional studies.

The investigators will be responsible for analyzing the study data, and the analysts will be blinded to patients' group assignment during the execution of the study. For the purpose of the final analysis, the official clinical database will not be unblinded until medical/scientific review has been completed and the investigators have been assured that the data are complete.

Before performing any analysis, the distribution of all variables will be examined for appropriateness of distribution assumptions. Descriptive statistics will be summarized for all variables including demographics, duration of analgesia, VAS scores during rest and after surgery, time for 1st rescue analgesia, total dose of rescue analgesia received in 24 hrs and side effects. Mean ± SD will be reported for continuous variables and frequency (percentage) will be reported for discrete variables. Analysis of variance or Kruskal-Wallis test as appropriate will be used to analyze and compare the primary endpoint VAS among two groups as well as the secondary endpoints. Chi-square test or extended Fisher's exact test as appropriate will be used for the comparison of the incidence of chronic pain as well as other side effects. All analyses will be performed using SAS 9.3 (Cary, NC) and a p-value less than 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Simple or radical unilateral mastectomy with or without axillary lymph node dissection.
* American Society of Anesthesia (ASA) I, II and III

Exclusion Criteria:

* Morbid obesity (body mass index > 40 kg/m2);
* Renal insufficiency (creatinine > 2.0 mg/DL),
* Current chronic analgesic therapy (daily use > 4 weeks),
* History of opioid dependence, pregnancy.
* Allergy to local anesthetic
* Rash/infection at the area of injection
* Coagulation disorder
* Patients on anticoagulation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of SPB block vs thoracic PVB | 6 months
  Efficacy of SPB block vs thoracic PVB block as described by reduce post operative pain score and reduce requirement for Narcotics.

SECONDARY OUTCOMES:
Onset and duration of block | 6 months
  Onset and duration of block as described by the time when block performed to the time of onset of block and Dermatomal distribution of sensory loss (tested with ice)
Post-operative rescue analgesia | up to 24 hours
  Time for 1st rescue analgesia
Development of chronic incisional pain | 24 and 48 hours
  Total dose of rescue analgesia received during the first 24 and 48 hrs
Pain related assessment scores as described in the Pain Detect Questionnaire | 6 months
  Pain related assessment scores as described in the Pain Detect Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sara Guzman-Reyes, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No